CLINICAL TRIAL: NCT04230759
Title: Radiochemotherapy +/- Durvalumab for Locally-advanced Anal Carcinoma.
Brief Title: Radiochemotherapy +/- Durvalumab for Locally-advanced Anal Carcinoma. a Multicenter, Randomized, Phase II Trial of the German Anal Cancer Study Group
Acronym: RADIANCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Daniel Martin, PD MD, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADIANCE; 2018-003005-25 (EudraCT Number); 70113615 (Other Grant/Funding Number: DKH); ESR-17-13077 (Other Grant/Funding Number: AstraZeneca); 2024-513914-36-00 (EU CTIS Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anal Cancer; Anal Carcinoma; Anal Cancer Stage III; Anal Cancer Stage II
Keywords: Anal Cancer; Anal Carcinoma; Durvalumab; PD-L1 immune checkpoint inhibitor
MeSH Terms: conditions — Anus Neoplasms | interventions — Drug Therapy; Fluorouracil; Radiation; durvalumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5FU+Mitomycin C (Active Comparator): Radiochemotherapy for anal cancer
  Interventions: Drug: Chemotherapy; Radiation: Radiation
- 5FU+Mitomycin C+Durvalumab (Experimental): Radiochemotherapy with Durvalumab for anal cancer
  Interventions: Drug: Chemotherapy; Radiation: Radiation; Drug: Durvalumab

INTERVENTIONS:
Drug: Chemotherapy — Patients receive chemotherapy cycles as followed:
  Mitomycin-C 12 mg/m², day 1 (maximum single dose 20 mg) 5-FU: 1000 mg/m² per day, continuous i.v. infusion, on day 1-4 and 29-32
  Other Names: all brands of 5-fluorouracil (5-FU) are allowed; all brands of Mitomycin C (MMC) are allowed
Radiation: Radiation — PTV_A (primary tumor): T1-T2<4cm N+: 28 x 1.9 Gy=53.2 Gy, five fractions per week or PTV_A (primary tumor): T2>=4cm, T3-4 Nany: 31 x 1.9 Gy=58.9 Gy, five fractions per week PTV_N (involved node): 28 x 1.8 Gy=50.4 Gy, five fractions per weeks PTV_Elec (elective node): 28 x 1.43 Gy=40.0 Gy, five fractions per week
Drug: Durvalumab — 1500 mg, 1h-civ, every 4 weeks (q4w) applied on day -14 (that is 14 days prior to initiation of RCT), day 15 (during RCT), and thereafter q4w (+/- 3d) for a total of 12 doses
  Other Names: PD-L1 inhibitor
  Arms: 5FU+Mitomycin C+Durvalumab

SUMMARY:
The RADIANCE multicenter, randomized phase II trial will assess the efficacy of durvalumab, a PD-L1 immune checkpoint inhibitor, in combination with primary mitomycin C (MMC)/5-fluorouracil (5-FU)-based radiochemotherapy (RCT) in patients with locally-advanced anal squamous cell carcinoma (ASCC).

DETAILED DESCRIPTION:
Anal squamous cell carcinomas (ASCC) are increasing in frequency across the developed world. There is a strong rationale for combining the PD-L1 immune checkpoint inhibitor durvalumab with radiochemotherapy (RCT) in patients with ASCC. First, although primary RCT with concurrent mitomycin C and 5-fluorouracil (MMC/5-FU) is the standard treatment for ASCC, the 3-year DFS in patients with locally-advanced disease is only in the range of 60%. Second, approximately 80-90% of patients with ASCC are human papilloma virus (HPV)-positive, which is associated with higher tumor "immunogenicity" in this malignancy that is known to correlate with better response to RCT as well as PD-1/PD-L1 immune checkpoint inhibitors. Also, PD-L1 expression was observed in 33%-62% of patients with locally advanced non-metastatic ASCC that correlated with tumor stage. Third, inhibition of the PD-1/PD-L1 axis showed encouraging responses in recurrent/metastatic ASCC in two phase Ib/II trials. Fourth, several data indicate complementary roles between R(C)T and immunotherapy. Fifth, R(C)T can induce PD-L1 upregulation with resulting dysfunction in CD8+ T-cells, and addition of anti-PD-L1 to R(C)T can overcome T-cell suppression to reinvigorate immune surveillance. First clinical studies have demonstrated promising findings for the combination of RCT and immunotherapies. Thus, based on the above data, RCT combined with durvalumab is expected to be more effective than primary RCT alone. Altogether, the hereby proposed RADIANCE multicenter, randomized phase II trial aims to improve the current standard treatment by incorporating durvalumab to the primary MMC/5-FU-based RCT in patients with locally-advanced ASCC (T2=>4cm Nany, stage IIB-IIIC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed ASCC (both genders) of the anal canal or the anal margin
* UICC-Stage IIB-IIIC including T2>4cm Nany (IIB: T3N0M0; IIIA: T1-2N1M0; IIIB: T4N0M0; IIIC: T3-4N1M0; T2>4cm Nany) according to proctoscopy, pelvic MRI, CT scan of thorax and abdomen, all within 30 days prior to recruitment
* Age ≥ 18 years, no upper age limit
* ECOG-Performance score 0-1
* History/physical examination within 30 days prior to recruitment
* Written informed consent and any locally-required authorization (e.g. EU Data Privacy Directive in the EU) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations
* Life expectancy of > 12 months
* Body weight >30kg
* Hemoglobin ≥9.0 g/dl
* Leukocytes >3.5 x 10 ^9/l
* Absolute neutrophil count (ANC) 1.5 x 10 9/l (> 1500 per mm3)
* Platelet count ≥100 x 109/l (>100,000 per mm3)
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT), ALT (SGPT), AP ≤ 3x institutional ULN
* Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula creatinine clearance
* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of durvalumab. A highly sensitive pregnancy test must be used.
* Female subjects of childbearing potential must be willing to use a highly effective contraceptive measure as defined in the Clinical Trial Facilitation Group (CTFG) guideline ("Recommendations related to contraception and pregnancy testing in clinical trials"). Highly effective contraception is required from screening to 90 days after the last dose of durvalumab. (Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.)
* Male subjects of childbearing potential must agree to use a highly effective method of contraception, starting from screening to 90 days after the last dose of durvalumab. (Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.) Male patients should refrain from fathering a child or donating sperm during the study and for 180 days after the last dose of durvalumab + any drug combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* For HIV-positive patients: running combined antiretroviral therapy (CART) on a stable dose at study entry and undetectable HIV-viral load (HIV Viral load <50 copies/mL and CD4>200/mircoliter). Patients will be closely monitored and CART management will be performed according to appropriate labelling guidance of the antiviral therapy. CART should be on a stable dose at study entry.

Exclusion Criteria:

* UICC-Stage I-IIA ASCC defined as cT1N0M0 or cT2 <4cm N0M0 disease
* Second malignancy other than basalioma or cervical/genital/ neoplasia in situ
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of durvalumab and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Known DPD-deficiency
* Participation in another clinical study with an investigational product during the last 12 months
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Any previous treatment with other immunotherapy, a PD1 or PD-L1 inhibitor
* QT interval corrected for heart rate (QTc) ≥470 ms
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/d of prednisone, or an equivalent corticosteroid. In case of recent introduction of CART, inclusion will be possible provided subjects had at least 4 weeks of treatment prior to inclusion.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Chairman.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Chairman
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment, other than the study medication. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Previous radiotherapy treatment to the pelvis or radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of durvalumab.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study chairman
  * Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of leptomeningeal carcinomatosis or any other metastatic disease
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab. Note: Patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and up to 30 days after the last dose of durvalumab.
* Known allergy or hypersensitivity to any of the study/investigational drugs or any of the study/investigational drug excipients and/or radiochemotherapy with 5-FU and Mitomycin C.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  DFS is defined as the time between randomization and the first of the following events: (a) non-complete clinical response at restaging MRI and proctoscopy, including biopsies of suspicious findings, 26 weeks after initiation of radiochemotherapy, (b) locoregional recurrence after initial complete clinical response (cCR), (c) distant metastases, (d) second primary cancer, or (e) death from any cause, whichever occurs first. Patients without any of these events are censored at the time point of last observation.

SECONDARY OUTCOMES:
Major adverse events | 3 Years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
cCR | 26 weeks
  Complete clinical response rate assessed 26 weeks after initiation of radiochemotherapy
Overall survival | 3 Years
  Overall survival defined as the time between randomization and death from any cause
Colostomy-free survival | 3 Years
  Colostomy-free survival defined as time between randomization and a definitive colostomy for progression, relapse, or complication
Cumulative incidence of locoregional recurrence | 3 Years
  Cumulative incidence of locoregional recurrence defined as the incidence of locoregional recurrence form the time of randomization
Cumulative incidence of distant recurrence | 3 Years
  Cumulative incidence of distant recurrence defined as the incidence of distant recurrence form the time of randomization
Quality of life questionnaires | 3 Years
  Quality of life questionnaire QLQ-C30
Quality of life questionnaires | 3 Years
  Quality of life questionnaire QLQ-ANL27

CONTACTS AND LOCATIONS:
Locations (25):
- Univeritätsklinik für Strahlentherapie-Radioonkologie, Graz, Austria
- Germany (23):
  - Institut für Radioonkologie und Strahlentherapie, Darmstadt, Darmstadt
  - Klinik und Poliklinik für Strahlentherapie und Radioonkologie, Dresden, Dresden
  - Klinik für Strahlenheilkunde, Universitätsklinikum Freiburg, Freiburg im Breisgau, Freiburg
  - Klinik und Poliklinik für Strahlentherapie, Essen, Hesse
  - UKSH Campus Kiel, Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig, Leipzig
  - Universitätsklinikum Magdeburg, Magdeburg, Magdeburg
  - Universitätsmedizin Mainz, Mainz, Mainz
  - Uniklinikum Marburg, Marburg, Marburg
  - Kliniken Maria Hilf GmbH Mönchengladbach, Mönchengladbach, Mönchengladbach
  - LMU Klinikum der Universität München, München, München
  - Technische Universität München, München, München
  - Universitätsklinikum Regensburg, Regensburg, Regensburg
  - Universitätsklinikum Rostock, Rostock, Rostock
  - Radioonkologie und Strahlentherapie, Berlin, State of Berlin
  - Universitätsklinik Tübingen, Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg, Würzburg
  - OnkoLibri GbR, Berlin
  - University Hospital Goethe University Frankfurt, Frankfurt
  - Universitätsmedizin Göttingen, Goettigen
  - Asklepios Klinik Altona, Hamburg
  - Hospital Barmherzige Brüder, Regensburg
  - Klinikum Stuttgart, Stuttgart
- UniversitätsSpital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No